CLINICAL TRIAL: NCT00391508
Title: An Epidemiological Study of Peristomal Skin Problems in Patient With an Ostomy in Roskilde County
Brief Title: Skin Problems in Ostomy Patients: An Epidemiological Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Zealand University Hospital (Other)
Collaborators: Coloplast A/S (Industry)
Other Study IDs: Sept-HN-2003
Record Dates: First submitted 2006-10-23; First posted 2006-10-24 (Estimated); Last update posted 2006-10-24 (Estimated); Status verified 2006-10

CONDITIONS: Ostomy; Living in Roskilde County; Persons More Than 18 Years of Age; Willingness to Participate
Keywords: Ostomy; Peristomal skin; Skin complication

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
Peristomal skin complications are thought to be common but the exact frequency and cause of these complications are unknown. We have sought to document the incidence of cutaneous peristomal problems and to find risk factors that might contribute to peristomal complications.

DETAILED DESCRIPTION:
Peristomal skin complications are thought to be common but the exact frequency and cause of these complications are unknown. We have sought to document the incidence of cutaneous peristomal problems and to find risk factors that might contribute to peristomal complications.

A cross sectional study was conducted from September 2003 to January 2005. The study population included all persons with an ostomy living in Roskilde County, Denmark. We have attempted to include all persons with an ostomy by contacting the local municipalities administering individual aid. Danish law (law of social service section 4 chapter 19 § 97) states that every person with a chronic disease is entitled to reimbursement for any aid needed. For ostomy patients this means that they are entitled to free stoma care products from selected merchants and without restriction to type or manufacturer of ostomy product. All ostomy patients are automatically enrolled in the database at the local municipality in order to received reimbursement for product cost. It was therefore assumed that all ostomy patients were registered, as the law provides benefits without restrictions, and self-payment for alternative purchases would involve substantial additional and unnecessary private expenditure for the individual ostomy patient.

A letter was sent to every ostomy patient by the municipalities, inviting them to participate. The ostomy patients willing to participate would then return the stamped and addressed envelope with their reply. For all patients who accepted the invitation, a physical examination was scheduled.

At the time of the examination a detailed registration form was filled out to provide standardised records of known risk factors and other data of possible pertinence to the investigation.

A careful physical examination was performed by a dermatologist, a stoma care nurse specialist and a resident. The majority of ostomy patients were seen at the dermatological department Roskilde University Hospital, but a few were seen at their homes due to advanced age or physical impairment. Personal details, medical histories, stoma appliances and daily stoma care routines were recorded along with a thorough examination of the peristomal area in regards to ostomy placemant, skin retraction, hernia, stoma height and width. A general skin examination was also undertaken. Each variable was recorded and further documented by colour photographs. To ensure that the participating patients correlated to the general population, a national computer based register of all ostomy patients in Denmark were compared to our patients in regards to ostomy type, sex, age and geographical location. Patients with a peristomal skin problem and a control (person without a skin problem) were selected from the cross-sectional study and invited for further examination. At this examination several non invasive test were conducted. These non invasive test included: D-squame tapes, Capacitans measurements , TEWL(transepidermal water loss) measurements , Tape stripping, Mecanical measurements of the skin and pH measurements.

ELIGIBILITY:
Inclusion Criteria:

* Ostomy
* Living in Roskilde County
* Persons more than 18 years of age
* Willingness to participate

Exclusion Criteria:

* Under 18 years of age
* Living outside Roskilde County
* If not able to comprehend the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2003-09; Study Completion 2005-08

CONTACTS AND LOCATIONS:
Overall Officials: Hanne Nybaek, MD, Principal Investigator — Dept. of Dermatology, Roskilde Hospital
Locations (1):
- Roskilde University Hospital, Dept. of Dermatology, Dk-4000 Roskilde, Denmark